CLINICAL TRIAL: NCT06103708
Title: Quantitative Perfusion Imaging of the Lower Limb in Peripheral Arterial Disease Using Contrast Enhanced Perfusion Ultrasound, Arterial Spin Labelling Magnetic Resonance Imaging and Perfusion Angiography
Brief Title: Quantitative Perfusion Imaging Using Contrast Enhanced Perfusion Ultrasound, MRI and Perfusion Angiography
Acronym: QPiPAD
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 145177
Record Dates: First submitted 2023-10-09; First posted 2023-10-27 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peripheral Arterial Disease is the narrowing and blocking of the blood vessels that supply the legs and feet. It is a common and progressive condition that affects patients of all backgrounds and genders and is more common in people with other problems such as heart disease, high blood pressure and diabetes mellitus as well being linked to ageing. It can be a severe disease and in 20% of patients can lead to pain on walking short distances and 2% of people can lead to painful ulceration, constant pain and can lead to amputation of part or all of the affected leg.

The investigators are researching 2 different types of new scanning techniques to measure the amount of blood that is circulating within the tissues of the leg and foot (known as tissue perfusion). The investigators want to measure tissue perfusion in people both with and without Peripheral Arterial Disease. This will help find a more sensitive method to diagnose Peripheral Arterial Disease earlier and help identify those with worsening arterial narrowing before they develop ulcers. Measuring tissue perfusion will guide doctors with decision about what procedure can be performed to improve blood flow in people with Peripheral Arterial Disease .

Patients with all degrees of Peripheral Arterial Disease will be eligible to take part in this study. The study will take part at University College London and Royal Free Hospital. The research will run along side normal investigations and treatment for Peripheral Arterial Disease and the study period will be 2 years.

Participants will undergo an ultrasound scan of the lower leg with an injection of a special dye into a vein in the arm, as well as a magnetic resonance

DETAILED DESCRIPTION:
Participants in this study will either be a group of healthy disease-free participants or participants with peripheral arterial disease.

In the Peripheral Arterial Disease group, participants care will not deviate from standard management and follow up protocols and their involvement in the study will require them to attend for additional scans for research purposes.

In order to formulate a research question and methodology the investigators have consulted international and local experts in tissue perfusion who use contrast enhanced ultrasound perfusion and Magnetic Resonance Imaging perfusion techniques. The methodology and research protocols have been developed with clinicians (Vascular surgeons, Interventional Radiologists and Clinical Vascular Scientists) experienced in caring for and treating patients with Peripheral Arterial Disease .

The published literature on tissue perfusion includes research in several organs including the brain, liver, kidneys and with limited but robust data on measuring perfusion in the tissues of the lower limb in people with Peripheral Arterial Disease . There is very limited data on comparing and contrasting the perfusion data produced from two different imaging techniques in the leg muscles within the same cohort. This is extremely important as there is currently no standardised and accepted marker for tissue perfusion to use as a benchmark. Therefore using two techniques will help validate the results.

Through this research a range of values of tissue perfusion will be produced that reflect health and different clinically assessed stages of Peripheral Arterial Disease , as well as provide objective evidence of improved tissue perfusion in patients undergoing routine revascularisation procedures to treat severe Peripheral Arterial Disease .

It is imperative to identify the range of normal tissue perfusion variables in participants without Peripheral Arterial Disease who are a similar age group to the participant disease cohort. This is important as prior research by other groups has identified potential age related reduction in tissue perfusion in patients without symptoms or diagnosed Peripheral Arterial Disease . Refining the tissue perfusion techniques in patients without Peripheral Arterial Disease , will provide invaluable repeatability testing with an aim to produce a reliably control data set with which the investigators can better understand the tissue perfusion deficits in patient with Peripheral Arterial Disease.

Further key choices in the investigator study design was the type of techniques chosen to measure tissue perfusion. On consultation with Patient groups the design of the study was paramount to not interfere with participants normal investigation and treatment for Peripheral Arterial Disease. The scan techniques the investigators propose to investigate can both by carried out as an adjunct to the routine imaging techniques used in the diagnosis and management of Peripheral Arterial Disease as recommended by National Guidelines.

The number of recruited healthy volunteers will be limited by careful consideration of power calculations based on the published literature. The clinicians caring for patients with Peripheral Arterial Disease will also be responsible for recruitment of participants.

The recruitment material will not make any therapeutic promises rather explain the nature of the study which is to help develop new scanning techniques. All patients under the care of vascular surgery who are undergoing scans to diagnose of manage their condition can potentially be included. Consenting of participants will be carried out by surgeons and interventional radiologists with prior research recruitment experience and who are fully aware of the ethical principles underpinning valid informed consent.

Participants will not be allocated to different treatment groups, however participants in this study will be recruited to reflect a range of clinical severity of Peripheral Arterial Disease . This research will be carried out in tandem to their routine outpatient clinic appointments and scans. The investigators have considered that research may lead to additional waiting or travel times being incurred to participants and therefore the protocol has been designed to perform both the contrast enhanced ultrasound and magnetic resonance imaging scan on the same day in geographically close proximity, in order to limit travel and delays.

Risks to participants will be mitigated by thorough and robust screening processes. Examples will include standardised magnetic resonance imaging safety questionnaires to ensure safety of the scan and echocardiogram to identify any patients with cardiac shunts that are a contraindication for contrast ultrasound scans.

In order to prevent any conflict of interest occurring the research group will be well integrated into the clinical team caring for patients. At the end of the study patients who have participated will continue to be monitored with routine scanning techniques as per national guidelines. All results will be shared with patients. In individuals where the study results show tissue perfusion deficits, any relevant data that may benefit their clinical care will be considered by the clinicians caring for them. This may include closer monitoring of their condition for instance.

In order to correlate tissue perfusion findings with clinical symptoms and outcomes, participants' medical notes will be reviewed. All data collected will be anonymised both during analysis and in publication or presentation.

ELIGIBILITY:
Inclusion Criteria:

Disease-free participants:

1. Adult patients older than 40 years old
2. Subjects able to and willing to give informed consent
3. Staff from University College London Hospital/University College London

Participants with Peripheral Arterial Disease :

1. Patients able to and willing to give informed consent
2. Peripheral Arterial Disease Rutherford Classification stages 1- 6
3. Patients referred by University College London Hospital or Royal Free Hospital.

Exclusion Criteria

Disease-free participants:

1. Prior history of Peripheral Arterial Disease
2. History of diabetes, tobacco smoking or cardiovascular, vasculitides or muscle disease
3. Any contraindication to magnetic resonance imaging or contrast enhanced ultrasound- metal implants not compatible with magnetic resonance imaging; documented allergy to SonoVue; patients with right-to-left shunts assessed with transthoracic echocardiogram, severe pulmonary hypertension (pulmonary artery pressure >90 mmHg), uncontrolled systemic hypertension, and in patients with adult respiratory distress syndrome and recent myocardial infarction/ acute coronary syndrome in the preceding 7 days.
4. Participants not from University College London Hospital/University College London

Peripheral Arterial Disease participants:

1. Concurrent and/or recent involvement in other research that is likely to interfere with the intervention within 3 months of study enrolment
2. Any contraindication to magnetic resonance imaging or contrast enhanced ultrasound - metal implants not compatible with magnetic resonance imaging; documented allergy to SonoVue; patients with right-to-left shunts assessed with transthoracic echocardiogram, severe pulmonary hypertension (pulmonary artery pressure >90 mmHg), uncontrolled systemic hypertension, and in patients with adult respiratory distress syndrome and recent myocardial infarction/ acute coronary syndrome in the preceding 7 days.
3. Patients outside University College London Hospital or Royal Free Hospital.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants for disease-free cohort will be recruited from University College London Hospital/University College London Participants with Peripheral Arterial Disease will be recruited directly by the clinical team at University College London Hospital or Royal Free Hospital.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
A novel quantitative imaging biomarker of tissue perfusion | 12 months
  A novel quantitative imaging biomarker of tissue perfusion will be measured as a reference value to guide clinical assessment in patients with peripheral arterial disease.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom